CLINICAL TRIAL: NCT03213691
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of Selumetinib (AZD6244 Hydrogen Sulfate) in Patients With Tumors Harboring Activating MAPK Pathway Mutations
Brief Title: Selumetinib Sulfate in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With Activating MAPK Pathway Mutations (A Pediatric MATCH Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01250; NCI-2017-01250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621E; APEC1621E (Other: Children's Oncology Group); APEC1621E (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Childhood Non-Hodgkin Lymphoma; Ann Arbor Stage IV Childhood Non-Hodgkin Lymphoma; Recurrent Childhood Central Nervous System Neoplasm; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Lymphoma, Non-Hodgkin | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib sulfate PO BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib; Drug: Selumetinib Sulfate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD 6244; AZD-6244; AZD6244; MEK Inhibitor AZD6244
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate

SUMMARY:
This phase II Pediatric MATCH trial studies how well selumetinib sulfate works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with MAPK pathway activation mutations that have spread to other places in the body and have come back or do not respond to treatment. Selumetinib sulfate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with selumetinib (AZD6244 hydrogen sulfate) with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor activating genetic alterations in the MAPK pathway.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with selumetinib (AZD6244 hydrogen sulfate) with advanced solid tumors (including CNS tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor MAPK activation mutations.

II. To obtain additional information about the tolerability of selumetinib (AZD6244 hydrogen sulfate) in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate other biomarkers as predictors of response to selumetinib (AZD6244 hydrogen sulfate) and specifically, whether tumors that harbor different mutations or fusions will demonstrate differential response to selumetinib (AZD6244 hydrogen sulfate) treatment.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive selumetinib sulfate 25 mg/m2/dose orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to molecular analysis for therapy choice (MATCH) to APEC1621E based on the presence of an actionable mutation

  * Note: patients with BRAF V600 actionable mutations of interest (aMOIs) will be preferentially assigned to APEC1621G (vemurafenib) if that study is open and they are otherwise eligible for it
* Patients must have a body surface area >= 0.5 m^2 at enrollment
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have iobenguane (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) and visible on more than one slice

  * Note: the following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * X-ray therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation

    * Note: radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iodine I 131 metaiodobenzylguanidine [131I-MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to selumetinib (AZD6244 hydrogen sulfate)
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 within 7 days prior to enrollment
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) within 7 days prior to enrollment >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): male 0.6; female 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): male 0.8; female 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): male 1; female 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): male 1.2; female 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): male 1.5; female 1.4
  * Age: >= 16 years; maximum serum creatinine (mg/dL): male 1.7; female 1.4
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age within 7 days prior to enrollment
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; (for the purpose of this study, the ULN for SGPT is 45 U/L) within 7 days prior to enrollment
* Serum albumin >= 2 g/dL within 7 days prior to enrollment
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study within 7 days prior to enrollment
* A blood pressure (BP) =< the 95th percentile for age, height, and gender measured within 7 days prior to enrollment; please note that 3 serial blood pressures should be obtained and averaged to determine baseline BP; patients with hypertension controlled on antihypertensive medications will be allowed if otherwise eligible
* Serum triglyceride level =< 300 mg/dL within 7 days prior to enrollment
* Serum total cholesterol level =< 300 mg/dL within 7 days prior to enrollment
* Patients must be able to swallow intact capsules whole
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study because there is currently no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal; females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study treatment; males with sexual partners who are pregnant or who could become pregnant (ie, women of child-bearing potential) should use effective methods of contraception for 12 weeks after completing the study to avoid pregnancy and/or potential adverse effects on the developing embryo
* Concomitant medications

  * Corticosteroids: patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
  * CYP3A4 agents: patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible; strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study
  * CYP2C19 agents: patients who are currently receiving drugs that are strong CYP2C19 inducers (e.g., rifampin, ritonavir) or inhibitors (e.g.., fluoxetine, fluvoxamine, ticlopidine) are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients with known significant ophthalmologic conditions (uncontrolled glaucoma, history of retinal vein occlusion or retinal detachment, excluding patients with longstanding findings secondary to existing conditions) are not eligible
* Patients with low grade glioma are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl E Allen, Principal Investigator — Children's Oncology Group
Locations (110):
- United States (108):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Eckstein OS, Allen CE, Williams PM, Roy-Chowdhuri S, Patton DR, Coffey B, Reid JM, Piao J, Saguilig L, Alonzo TA, Berg SL, Ramirez NC, Jaju A, Mhlanga J, Fox E, Hawkins DS, Mooney MM, Takebe N, Tricoli JV, Janeway KA, Seibel NL, Parsons DW. Phase II Study of Selumetinib in Children and Young Adults With Tumors Harboring Activating Mitogen-Activated Protein Kinase Pathway Genetic Alterations: Arm E of the NCI-COG Pediatric MATCH Trial. J Clin Oncol. 2022 Jul 10;40(20):2235-2245. doi: 10.1200/JCO.21.02840. Epub 2022 Apr 1. PMID 35363510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Selumetinib)
Started | 21
Completed | 0
Not Completed | 21
Not completed — Adverse Event | 2
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 14
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: A responder is defined as a patient who achieves a best response of partial response (PR) or complete response (CR) on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors.
Time Frame: From enrollment to the end of treatment, up to 2 years
Population: One patient was deemed ineligible by the Study Chair and is excluded from this analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 20
Percentage of patients | 0

2. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events as Accessed by Common Terminology Criteria for Adverse Events (CTCAE) Version (v) 5.0
Description: A patient will be counted only once for a given toxicity for the worst grade of that toxicity reported for that patient.
Time Frame: From enrollment to the end of treatment, up to 2 years
Population: One patient was deemed ineligible by the Study Chair and is excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 20
Percentage of patients | 90 [68.3 to 98.8]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival will be defined as time from the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause. PFS along with the confidence intervals will be estimated using the Kaplan-Meier method.
Time Frame: From the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause, assessed up to 5 years
Population: One patient was deemed ineligible by the Study Chair and is excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 20
Percentage of patients | 15 [4.0 to 34.0]

4. Other Pre Specified Outcome: Biomarker Analysis as Predictors of Response to Selumetinib
Description: A descriptive analysis will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to 4.5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Tumor Genomic Profile
Description: as for outcome 4
Time Frame: Up to 4.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to 30 days after the end of treatment, up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Selumetinib)
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=20)
Papilledema (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ileal obstruction (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Disease progression (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
CPK increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hematoma (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=20)
Anemia (Blood and lymphatic system disorders) | 8
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Cushingoid (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Keratitis (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Retinopathy (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 7
Fever (General disorders) | 1
Gait disturbance (General disorders) | 2
Localized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Paronychia (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 2
Blood corticotrophin decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
CPK increased (Investigations) | 5
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 4
Ejection fraction decreased (Investigations) | 1
GGT increased (Investigations) | 1
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03213691/Prot_SAP_000.pdf